CLINICAL TRIAL: NCT07252115
Title: Multicenter Randomized Clinical Trial on the Efficacy and Safety of the Total Left-side Surgical Approach (TLSA) Versus the Traditional Bilateral Surgical Approach (TBSA) for Hiatal Hernia With Gastroesophageal Reflux Disease
Brief Title: TLSA Versus TBSA Surgical Approach for Hiatal Hernia With Gastroesophageal Reflux Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-P2-097-02
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: Hernia, Hiatal; GERD (Gastroesophageal Reflux Disease)
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic total left-sided surgical approach (Experimental)
  Interventions: Procedure: Laparoscopic total left-sided surgical approach
- Laparoscopic traditional bilateral approach (Active Comparator)
  Interventions: Procedure: Laparoscopic traditional bilateral approach

INTERVENTIONS:
Procedure: Laparoscopic total left-sided surgical approach — The intervention group adopts the laparoscopic complete left-sided surgical approach.
  Arms: laparoscopic total left-sided surgical approach
Procedure: Laparoscopic traditional bilateral approach — The control group adopts the laparoscopic bilateral surgical approach.
  Arms: Laparoscopic traditional bilateral approach

SUMMARY:
Gastroesophageal reflux disease (GERD), characterized by pathological reflux of gastric contents, affects 10%-20% of the global population with Western predominance and escalating incidence over recent decades. Anatomical and functional abnormalities of the esophagogastric junction (EGJ) such as hiatal hernia (HH) is one of the major pathophysiological mechanisms. GERD elevates risks for Barrett esophagus, esophageal adenocarcinoma and interstitial pulmonary fibrosis, while characteristic symptoms including reflux and heartburn substantially impair quality of life (QoL). Proton pump inhibitors (PPIs) are used to alleviate symptoms and prevent reflux-related esophageal mucosal damage, but may cause long-term adverse effects.

Anti-reflux surgery (ARS) is a well-established therapeutic option for patients with anatomical abnormalities, chronic PPI-refractory symptoms or unwilling to take lifelong PPIs. It provides comparable or potentially superior efficacy to PPIs, especially in reconstructing anatomical structures and addressing EGJ functional deficiencies. Maximize patients' QoL while minimizing side effects is priority for ARS. Despite advancements in surgical techniques, ARS remains invasive and is associated with inherent mechanical complications, including dysphagia and potential vagus nerve injury. A growing consensus recognizes that hepatic vagus nerve injury, occurring in a significant proportion of patients following ARS, potentially contributes to postoperative dysfunctions such as delayed gastric emptying, impaired reflux control, dyspeptic symptoms, cholelithiasis, ultimately diminishing QoL.

Although the traditional bilateral surgical approach (TBSA) is widely used, its requisite dissection of the lesser omentum invariably injures or severs the hepatic branch of the vagus nerve. The hepatic branch of the vagus arises from the anterior trunk and predominantly innervates the gastric antrum, pylorus, proximal duodenum and biliary tract. Functionally, it mediates a spectrum of vital physiological process including hepato-gastric reflexes that facilitate gastric motility via osmotic sensing, as well as glucose-sensitive reflexes that inhibit gastric motility and delay gastric emptying. Furthermore, hepatic branch is involved in food intake and metabolic homeostasis, and it exerts parasympathetic control over the coordinated contraction of the gallbladder and sphincter of Oddi. However, the functional preservation of the hepatic branch of the vagus nerve during ARS remains poorly understood, with limited clinical evidence and absent robust guidelines.

Based on our preliminary findings, we initiated a long-term evaluation of the total left-side approach (TLSA), a nerve-sparing strategy that preserves the lesser omentum and hepatogastric ligament to safeguard the hepatic branch of the vagus nerve, with the aim of enhancing postoperative QoL.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years.
* Confirmed diagnosis of hiatal hernia (type I to IV).
* Diagnosis of refractory GERD, defined as persistent symptoms despite receiving 40 mg daily omeprazole for 8-12 weeks.
* GERD confirmed by either:
* Increased esophageal acid exposure time (AET) on 24-hour pH monitoring, and/or
* Endoscopic evidence of esophagitis.
* Hiatal hernia diagnosis verified by both abdominal CT and gastroscopy.

Exclusion Criteria:

* Presence of GERD without a hiatal hernia.
* Esophageal motility disorder.
* History of esophageal or other upper abdominal surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Quality of Life Index (GLQI) | Follow-up begins after surgery, with each patient followed for 3 years at the following time points: 3, 6, 12, 18, 24, and 36 months. Questionnaire surveys are completed at each time point.
  GIQLI is related to the QOL for gastrointestinal disorders. It contains 5 subscales, with a score range of 0 to 144 points. The higher the score, the better the patient's QOL and the better the surgical effect.

SECONDARY OUTCOMES:
esophagitis | 1 and 3 years after surgery
  varified by gastroscopy （LA-standard）
DeMeester score | 1 and 3 years after surgery
  The DeMeester score is a quantitative index used to distinguish between pathological and physiological acid reflux. It is calculated as a composite score based on multiple parameters derived from 24-hour esophageal pH monitoring, primarily the percentage of time the esophageal pH falls below a threshold of 4. A score greater than 14.7 is indicative of pathological acid reflux, whereas a score below this threshold is considered within the physiological range.
Incidence of gallstones | postoperative 1 and 3-year
  abdominal ultrasonography
Gastrointestinal Symptom Rating Scale | Follow-up begins after surgery, with each patient followed for 3 years at the following time points: 3, 6, 12, 18, 24, and 36 months. Questionnaire surveys are completed at each time point.
  The GSRS comprises 15 items, encompassing five symptom domains: Abdominal Pain Syndrome, Indigestion Syndrome, Diarrhea Syndrome, Constipation Syndrome, and Reflux Syndrome. Each item is rated on a 7-point Likert scale (where 1 represents "no symptoms" and 7 represents "very severe symptoms"). Each symptom item is scored individually (1-7), resulting in a total score range of 15 to 105. Higher total or domain scores indicate more pronounced symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided